CLINICAL TRIAL: NCT04405869
Title: Incidence of Thromboembolic Events and Prognosis of COVID-19 Patients Hospitalized in Intensive Care Units in France
Brief Title: Thromboembolic Events in Severe COVID-19 Patients
Acronym: COVICLOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7779
Record Dates: First submitted 2020-05-25; First posted 2020-05-28 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Pulmonary Thromboembolism
Keywords: Covid-19; Thrombosis; D-Dimers; Anticoagulation
MeSH Terms: conditions — Pulmonary Embolism; COVID-19; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of this study is to describe the incidence of thromboembolic events in a population of patients hospitalized in intensive care units in France for severe COVID-19. The secondary objective of this study is to describe the evolution of hemostasis parameters during the first two weeks of intensive care hospitalization and to evaluate the influence of different anticoagulation regimens on these parameters and on the incidence of thromboembolic events

ELIGIBILITY:
Inclusion Criteria:

* Confirmed infection with the Sars-CoV-2 virus (RT-PCR)
* Hospitalization in Intensive Care Unit
* Age over 18 years Old

Exclusion Criteria:

* Refusal of the patient to participate in data collection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed infection with the Sars-CoV-2 virus
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Analysis of incidence of thromboembolic events in patients with Sars-CoV-2 | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie-Réanimation - Nouvel Hôpital Civil, Strasbourg, France

REFERENCES:
- [Derived] Tacquard C, Mansour A, Godon A, Godet J, Poissy J, Garrigue D, Kipnis E, Rym Hamada S, Mertes PM, Steib A, Ulliel-Roche M, Bouhemad B, Nguyen M, Reizine F, Gouin-Thibault I, Besse MC, Collercandy N, Mankikian S, Levy JH, Gruel Y, Albaladejo P, Susen S, Godier A; French Working Group on Perioperative Hemostasis. Impact of High-Dose Prophylactic Anticoagulation in Critically Ill Patients With COVID-19 Pneumonia. Chest. 2021 Jun;159(6):2417-2427. doi: 10.1016/j.chest.2021.01.017. Epub 2021 Jan 16. PMID 33465342